CLINICAL TRIAL: NCT02145871
Title: A Prospective Randomized Controlled Clinical Trial of Standard Versus Goal-Directed Perioperative Fluid Management (GDT) for Patients Undergoing Radical Cystectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-069
Record Dates: First submitted 2014-05-21; First posted 2014-05-23 (Estimated); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Bladder Cancer
Keywords: Radical Cystectomy; Perioperative Fluid Management; EV1000; 14-069
MeSH Terms: conditions — Urinary Bladder Neoplasms

ARMS (2):
- Standard fluid management (Active Comparator): The non-intervention group will receive maintenance crystalloid fluid at 10cc/kg/h. Blood loss will be replaced 1:1 with albumin. Transfusion will follow transfusion criteria. Fluid management will not be dependent on the EV1000
  Interventions: Other: standard fluid management
- Goal directed fluid therapy (GDT) (Experimental): In the GDT arm, patient's SV will be optimized before induction with crystalloid boluses prior to induction of general anesthesia. The GDT arm will have fluid therapy guided by the Edwards EV1000-clinical platform and maintenance crystalloid fluid will be 3cc/kg/h. During the surgical procedure when SVV rises above 12 an albumin bolus will be administered at 250 ml increments until the SVV falls below 8. Transfusion will follow transfusion criteria.
  Interventions: Other: fluid management guided by the EV1000

INTERVENTIONS:
Other: standard fluid management
  Arms: Standard fluid management
Other: fluid management guided by the EV1000
  Arms: Goal directed fluid therapy (GDT)

SUMMARY:
The purpose of this study is to help us learn what is the best amount of fluid to give to patients during bladder surgery in order to avoid delayed bowel function after surgery, which could prolong hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Adults (21 years old or greater) who are able to provide informed consent
* Patients who undergo an open, elective radical cystectomy

Exclusion Criteria:

* Patients with active atrial fibrillation or flutter, since the algorithm is not accurate in case of cardiac arrhythmia
* Female patients who are pregnant (female patients of child-bearing potential must have a negative serum pregnancy test ≤ 14 days prior to surgery or 15 to 30 days prior to surgery with a negative urine pregnancy test the morning of surgery)
* Presence of ascites, because increased abdominal pressure interferes with EV1000 reading accuracy
* BMI > 45 or <17, because increased abdominal pressure interferes with EV1000 reading accuracy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2014-05-21 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-03-14 (Actual)

PRIMARY OUTCOMES:
incidence of postoperative ileus (POI) | 3 years
  POI will be defined as intolerance of oral intake by postoperative day 5, or the cessation of diet and/or placement of an NGT for clinical signs or symptoms associated with POI, including one or more of the following: nausea, emesis, abdominal bloating or distension, or excessive burping. Rate of ileus will be compared between the treatment groups using the chi-square test. A 95% confidence interval for the difference in ileus rate will also be reported.

SECONDARY OUTCOMES:
complications | 1 year post operatively
  Overall rate of grade 2-5 1-year complications, and rate of grade 2-5 gastrointestinal, pulmonary, renal, hematologic and cardiac complications will also be compared using the chi-square test. Based rate of grade 2-5 gastrointestinal, pulmonary, renal, hematologic and cardiac complications will also be compared using the chi-square test.
compare total volume of fluid | the first 72 hours
  given intraoperatively and during the first 72 hrs postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Vittoria Arslan-Carlon, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/